CLINICAL TRIAL: NCT04390711
Title: An Observational Cross-sectional Study to Compare Carbamylated High-density Lipoprotein Levels Among Normal Subjects, Type 2 Diabetes Mellitus Patients With and Without Coronary Heart Disease.
Brief Title: Association of Carbamylated HDL and CAD in T2DM Patients
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: c-HDL study
Record Dates: First submitted 2020-05-08; First posted 2020-05-15 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus With Circulatory Complciation
Keywords: Carbamylation,HDL,T2DM

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subjects: We included 40 age- and gender-matched healthy subjects to serve as the control group, who had normal blood pressure, serum fasting glucose, lipid profile, and renal function.
  Interventions: Other: High density lipoprotein isolation, detection and in-vitro study.
- T2DM with CAD: Diagnosis of T2DM was made according to the criteria of the American Diabetes Association. All patients were tested by angiography, with CAD diagnosed if luminal diameter narrowing was estimated visually at ≥50% in a major epicardial coronary artery.
  Interventions: Other: High density lipoprotein isolation, detection and in-vitro study.
- T2DM without CAD: Diagnosis of T2DM was made according to the criteria of the American Diabetes Association.T2DM without CAD was diagnosed if no luminal diameter narrowing was estimated visually at ≥50% in a major epicardial coronary artery.
  Interventions: Other: High density lipoprotein isolation, detection and in-vitro study.

INTERVENTIONS:
Other: High density lipoprotein isolation, detection and in-vitro study. — All blood samples were taken on the day of cardiac catheterization after overnight fasting.High density lipoprotein from each participants was isolated and further collected for carbamylation level detection and in-vitro study.

SUMMARY:
This is an observational cross-sectional study aimed at investigating the alterations of the carbamylated-HDL levels in T2DM patients, and comparing the concentration of carbamylated-HDL between the T2DM patients with CAD and without CAD to explore the association between carbamylated-HDL and risk of CAD in T2DM patients.

DETAILED DESCRIPTION:
High-density lipoprotein (HDL) is involved in various atheroprotective processes, including reverse cholesterol transport, inhibition of lipid oxidation and inflammatory cytokine secretion, endothelial repair, and antiapoptotic function, which all contribute to the regression of plague burden. Recent studies have shown that oxidative stress and chronic inflammation - both implicated in the process of diabetes - can contribute to an irreversible post-translational modification called carbamylation. Carbamylation levels reflect the burden of enhanced inflammation, oxidative stress, and renal impairment, and can serve as a biomarker of certain pathological conditions. Several clinical studies have demonstrated positive associations between cardiovascular risk, mortality, and serum carbamylation-derived product levels in the general population and particularly in patients with kidney failure. Increasing evidence also shows that carbamylated lipoprotein plays a pivotal role in atherosclerosis.18 However, most studies concerning carbamylation have been performed under a kidney disease background. Whether HDL particles in patients with type 2 diabetes mellitus (T2DM) show enhanced carbamylation and whether this enhancement is associated with vascular complications remains unknown. Thus, in the present study, the investigators aim to test whether HDL experiences carbamylation in T2DM patients and investigated the pro-atherogenic effects of carbamylated HDL on endothelial-monocyte adhesion.

ELIGIBILITY:
Inclusion Criteria:

1:Clinical diagnosis of T2DM (according to the criteria of the American Diabetes Association.)

Exclusion Criteria:

1. end-stage renal disease (ESRD)
2. acute coronary syndrome,
3. heart failure,
4. chronic viral or bacterial infection,
5. cancer,
6. immune system disorders

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between September 2018 to March 2019, a total of 242 consecutive T2DM patients who visited Shanghai Ruijin Hospital were enrolled in this study. All patients were tested by angiography, with CAD diagnosed if luminal diameter narrowing was estimated visually at ≥50% in a major epicardial coronary artery. Patients with end-stage renal disease (ESRD) (n = 9), acute coronary syndrome(n = 25), heart failure (n = 21), chronic viral or bacterial infection (n = 7), tumors(n = 8), or immune system disorders (n = 3) were excluded from this study. We included 40 age- and gender-matched healthy subjects to serve as the control group, who had normal blood pressure, serum fasting glucose, lipid profile, and renal function.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Carbamylated-HDL levels alteration between the control and the T2DM patients with and without concomitant CAD. | within 1week after enrollment
  HDL was isolated from subjects' plasma and its carbamylation levels were further detected by the enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, MD, Study Director — Department of Cardiology, Ren Ji Hospital
Locations (1):
- Rui Jin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenson RS, Brewer HB Jr, Ansell BJ, Barter P, Chapman MJ, Heinecke JW, Kontush A, Tall AR, Webb NR. Dysfunctional HDL and atherosclerotic cardiovascular disease. Nat Rev Cardiol. 2016 Jan;13(1):48-60. doi: 10.1038/nrcardio.2015.124. Epub 2015 Sep 1. PMID 26323267
- [Background] Sun JT, Liu Y, Lu L, Liu HJ, Shen WF, Yang K, Zhang RY. Diabetes-Invoked High-Density Lipoprotein and Its Association With Coronary Artery Disease in Patients With Type 2 Diabetes Mellitus. Am J Cardiol. 2016 Dec 1;118(11):1674-1679. doi: 10.1016/j.amjcard.2016.08.044. Epub 2016 Aug 30. PMID 27666175
- [Background] Femlak M, Gluba-Brzozka A, Cialkowska-Rysz A, Rysz J. The role and function of HDL in patients with diabetes mellitus and the related cardiovascular risk. Lipids Health Dis. 2017 Oct 30;16(1):207. doi: 10.1186/s12944-017-0594-3. PMID 29084567
- [Background] Delanghe S, Delanghe JR, Speeckaert R, Van Biesen W, Speeckaert MM. Mechanisms and consequences of carbamoylation. Nat Rev Nephrol. 2017 Sep;13(9):580-593. doi: 10.1038/nrneph.2017.103. Epub 2017 Jul 31. PMID 28757635
- [Background] Sun JT, Yang K, Mao JY, Shen WF, Lu L, Wu QH, Wang YP, Wu LP, Zhang RY. Cyanate-Impaired Angiogenesis: Association With Poor Coronary Collateral Growth in Patients With Stable Angina and Chronic Total Occlusion. J Am Heart Assoc. 2016 Dec 16;5(12):e004700. doi: 10.1161/JAHA.116.004700. PMID 27986757
- [Background] Long J, Vela Parada X, Kalim S. Protein Carbamylation in Chronic Kidney Disease and Dialysis. Adv Clin Chem. 2018;87:37-67. doi: 10.1016/bs.acc.2018.07.002. Epub 2018 Aug 23. PMID 30342712
- [Background] Verbrugge FH, Tang WH, Hazen SL. Protein carbamylation and cardiovascular disease. Kidney Int. 2015 Sep;88(3):474-8. doi: 10.1038/ki.2015.166. Epub 2015 Jun 10. PMID 26061545
- [Derived] Chen Z, Ding S, Wang YP, Chen L, Mao JY, Yang Y, Sun JT, Yang K. Association of carbamylated high-density lipoprotein with coronary artery disease in type 2 diabetes mellitus: carbamylated high-density lipoprotein of patients promotes monocyte adhesion. J Transl Med. 2020 Dec 3;18(1):460. doi: 10.1186/s12967-020-02623-2. PMID 33272295